CLINICAL TRIAL: NCT05274334
Title: Measurement of Lipogenic Flux by Deuterium Resolved Mass Spectrometry Via Non-invasive Breath Analysis
Acronym: D2OBREATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Swiss National Science Foundation (Other); Fondation Botnar (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-00099; ks22Sinues
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: De Novo Lipogenesis (DNL)
Keywords: deuterium resolved mass spectrometry; exhaled breath; deuterium enrichment; metabolome of exhaled breath; deuterated exhaled metabolites

STUDY DESIGN:
Intervention Model Description: One arm, Proof of Concept Study assessing metabolites in exhaled breath of healthy adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): Assessment of de novo lipogenesis non-invasively in exhaled breath in overnight-fasted humans by triggering feeding response by deuterium resolved mass spectrometry.
  Interventions: Other: Assessment of de novo lipogenesis non-invasively in exhaled breath

INTERVENTIONS:
Other: Assessment of de novo lipogenesis non-invasively in exhaled breath — 1. Healthy participants have a good nights sleep whereas they don't eat during the night and until measurements.
  2. They come to the lab and make first baseline exhalation sets. An exhalation set consists of 6 exhalations in Mass Spectrometer positive mode and the same in negative mode. One exhalation set takes around 7minutes from start to finish.
  3. Participants consume a single oral dose of dose of 70% 2H2O at 2 g/kg body-water.
  4. Participants execute several exhalation sets over time.
  5. Participants consume 300g of 'Excellence Joghurt Nature gezuckert.
  6. Participants execute several exhalation sets over time.
  7. After around 4.5hours with regular exhalation sets taking place, the trial is concluded.

SUMMARY:
This proof of concept- study is to measure de novo lipogenesis (DNL) non-invasively in exhaled breath in overnight-fasted humans by triggering feeding response by deuterium resolved mass spectrometry.

DETAILED DESCRIPTION:
The study objective is to measure the DNL by ingestion of a single oral dose of 70% 2H2O at 2 g/kg body-water. The subjects will consume a Yoghurt consisting of 300g of 'Excellence Joghurt Nature gezuckert' which contains 410 Kcal, 28g fat, 34g carbohydrates and 9g protein. The exhaled air of the subjects will be measured several times per hour to analyse de novo lipogenesis (DNL) non-invasive by deuterium resolved mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers
* English speaking, or good knowledge of the English language
* Able to understand the study
* Able to give informed consent

Exclusion Criteria:

* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Variation of signal intensity of deuterated exhaled metabolites across the approximately lasting 4.5 hours trial | approximately 4.5 hours
  Variation of signal intensity of deuterated exhaled metabolites across the approximately lasting 4.5 hours trial

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Sinues, Prof. Dr., Principal Investigator — Universitäts-Kinderspital beider Basel (UKBB)
Locations (1):
- University Children's Hospital Basel (UKBB), Basel, Switzerland